CLINICAL TRIAL: NCT06364527
Title: Use of Aptar Digital Health's Respiratory Disease Management Platform for Asthma: A Pilot Study
Brief Title: Use of Aptar Digital Health's Respiratory Disease Management Platform for Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CoheroHealth (Industry)
Collaborators: Aptar Digital Health (Industry); Lindus Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ADH-BSA-02-23
Record Dates: First submitted 2024-03-27; First posted 2024-04-15 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Asthma Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with fractioned exhaled nitric oxide ≥ 45 ppb (Experimental): Group 1 consists of 59 participants with a fractioned exhaled nitric oxide ≥ 45 ppb and ≥ 3 exacerbations / year (biologic eligible). Group 2 consists of 59 participants with a fractioned exhaled nitric oxide ≥ 45 ppb and < 3 exacerbations / year (biologic ineligible).
  Interventions: Device: Aptar Digital Health respiratory disease management platform

INTERVENTIONS:
Device: Aptar Digital Health respiratory disease management platform — The Aptar Digital Health respiratory disease management platform is a digital health tool that combines a Healthcare Professional portal (BreatheSmart Connect) and an associated patient mobile application (BreatheSmart mobile application). The Aptar Digital Health respiratory disease management platform is intended to be used in conjunction with compatible connected sensor devices that track medication adherence and for some, technique.

SUMMARY:
The United Kingdom has a high prevalence of asthma (over 12%) and some of the worst health outcomes in Europe. The management of respiratory disease and associated patient outcomes has long been an area of focus and improvement for the National Health Service. With the advancement of digital health technology, there is the potential to transform patient care and improve outcomes.

The Aptar Digital Health respiratory disease management platform, a digital therapeutic will be utilized to determine its value and how it supports: i) asthma patient engagement and facilitates communication between patients and providers to accelerate medication adherence; ii) asthma control through the use of the Asthma Control Questionnaire-5. In addition, spirometry and fractioned exhaled nitric oxide will be utilized during the study to validate and enhance current National Institute for Health and Care Excellence guidelines.

DETAILED DESCRIPTION:
This is an open-label, single comparative study that will accrue a total of 118 participants and compare pre and post study results. Group # 1 will consist of 59 participants with a fractioned exhaled nitric oxide ≥ 45 ppb and ≥ 3 exacerbations / year (biologic eligible). Group # 2 will consist of 59 participants with a fractioned exhaled nitric oxide ≥ 45 ppb and < 3 exacerbations / year (non-biologic eligible). At the baseline visit, clinic appointment # 1, health care providers will review the participants' medical records to determine clinical outcomes in the past year, including number of exacerbations, medication pharmacy refill percentage, and fractioned exhaled nitric oxide score. At the baseline visit, participants will also complete the Asthma Control Questionnaire-5 and the Mini-Asthma Quality of Life Questionnaire. The past year clinical evaluation and Asthma Control Questionnaire-5 and Mini-Asthma Quality of Life Questionnaire will be considered baseline results.

Patients will be screened for study appropriateness at the Guy's Hospital Severe Asthma Clinic. During the initial visit, which will be considered the study baseline visit, patients will be provided with the Aptar Digital Health respiratory disease management platform and trained to use the platform. Participants will be scheduled for in person follow-up visits at 1-2 months and then 6-months post-baseline; patients will be scheduled for virtual visits at 3-months post-baseline.

Patients will then be trained by Guy's Hospital team members; Aptar Digital Health staff will provide extensive training to the Guy's Hospital team prior to the study to ensure the team is fully knowledgeable about the product, its features, and can successfully onboard participants onto the Aptar Digital Health respiratory disease management platform. Once participants are trained, they will utilize the BreatheSmart mobile application by downloading it through either the Apple Store™ or Google Play™.

The BreatheSmart mobile application records, stores, and transmits usage events to the HeroTracker sensors, or via manual user entry, to a remote storage system. Participants may self-enter their medication schedule either with or without the help of their health care providers. Through the BreatheSmart mobile application, they can review information collected from the HeroTracker Sense metered dose inhaler and FindAir ONE dry powder inhaler sensors, report and review their adherence and self-reported symptoms, and answer validated questionnaires.

Participants can share the data entered through the BreatheSmart mobile application with caregivers and health care providers. Health care providers are then able to utilize BreatheSmart Connect, a web application, to obtain an overview of all participants utilizing the Aptar Digital Health respiratory disease management platform including detailed views of individual participant information. Health care providers can view real-time adherence, medication list, participants within and outside of risk zones (depending on adherence), rescue medication usage, symptoms, and triggers. Based on the information gleaned from the BreatheSmart Connect platform, clinicians will schedule follow-up participant appointments with either a junior or senior pharmacist at the Guy's Hospital Severe Asthma Clinic.

Participants will use the Aptar Digital Health respiratory disease management platform for 6 months and will be required to return the device upon study completion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years
* Utilization of asthma controller therapy: inhaled corticosteroids (ICS), long-acting β2-agonists (LABAs) and/or fixed combination therapies of LABA and ICS (medium to high-dose ICS/LABA therapy)
* Use of metered dose inhaler (MDI) and / or dry powder dose inhaler (DPI) list of compatible medications is noted in section 9.2.
* FeNO ≥ 45 ppb
* Primary respiratory diagnosis of asthma
* Patients with uncontrolled, moderate-to-severe asthma
* Non-smoker
* Capable of giving signed informed consent, which includes compliance with requirements and restrictions listed in consent form and protocol.
* Subject understands and is willing, able, and likely to comply with study procedures and restrictions
* Willingness to participate in this study and to use the Aptar Digital Health technology
* Willingness to share information / data with Aptar Digital Health (through informed consent)

Access to technology

* Access to a smartphone (requirements Android ≥13 and iOS ≥16
* Ability to use smartphone (smartphone usability assessment to be provided by Aptar Digital Health)
* Access to a current email account
* Access to data / Wi-Fi

Exclusion Criteria:

* Age < 16 years
* FeNO < 45 ppb
* Known or suspected alcohol or drug abuse which in opinion of investigator could interfere with subject's proper completion of the protocol requirement
* History of life-threatening asthma: Defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within last 6 months
* A lower respiratory tract infection within 7 days of the screening visit
* Concurrent diagnosis of chronic obstructive pulmonary disease (COPD) or other respiratory disorders including active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases.
* History of hypersensitivity/intolerance to any components of the study inhalers (example, lactose, magnesium stearate). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates participation will also be excluded.
* Ever received treatment with biological based therapy example, omalizumab, mepolizumab, for asthma.
* Received an investigational drug and/or medical device within 30 days of entry into this study (Screening), or within five drug half-lives of the investigational drug, whichever is longer
* An immediate family member of the participating investigator, sub-investigator, study coordinator, employee of the participating investigator, or any family member of a Aptar Pharma, Aptar Digital Health, Voluntis, or Cohero employee.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Questionnaire - 5 scores | 6 months
  Asthma Control Questionnaire - 5 has 5 questions each ranging from a low of 0 to a high of 6. 0 indicates "never" and 6 indicates "always". The minimum mean score is a 0 and the highest mean score is a 6. The lower the score the better the outcome.
  Change in normal distribution and mean Asthma Control Questionnaire - 5 scores from baseline to 6 months, which is the end of the study.

SECONDARY OUTCOMES:
Mini-Asthma Quality of Life Questionnaire | 6 months
  Mini-Asthma Quality of Life Questionnaire has 15 questions each ranging from a low of 1 to a high of 7. 1 indicates "all the time" and 7 indicates "none of the time". The higher the mean score the better the outcome.
  Change in normal distribution and mean values of Mini-Asthma Quality of Life Questionnaire scores from baseline to 6-months, which is the end of study.
Rescue medication usage | 6 months
  Asthmatics are prescribed two medications: 1) controller; 2) rescue. The controller medication schedule is prescribed by the healthcare provider. Rescue medication is used on an "as needed" basis when an asthmatic needs immediate relief due to an exacerbation.
  The lower the use of rescue medication, the better. The higher the use of rescue medication, the worse.
  Change in normal distribution and mean values of rescue medication usage (calculated on a daily and per patient basis) from baseline to 6-months, which is the end of study.
Inhaled corticosteroid steroid daily adherence | 6 months
  Asthmatics are prescribed two medications: 1) controller inhaled corticosteroid; 2) rescue. The controller inhaled corticosteroid steroid schedule is prescribed by the healthcare provider and is usually scheduled to be taken on a daily basis. If a patient is supposed to take their controller inhaled corticosteroid medication twice in one day and takes it twice, their adherence to their controller inhaled corticosteroid would be 100% on that day. If the patient is supposed to take it twice, but only takes it once, then their adherence to their controller inhaled corticosteroid would be 50% on that particular day.
  The higher the adherence the better the outcome. The lower the adherence the worse the outcome.
  Change in normal distribution and mean values of controller inhaled corticosteroids adherence from baseline to 6-months, which is the end of study.

OTHER OUTCOMES:
Step-up from inhaled corticosteroids to biologics | 6 months
  Some patients with severe asthma may require stronger medication, known as biologics, which are injectables. The thought is that if adherence and technique to a patient's controller inhaled corticosteroid can be improved, there could be a subset of severe patients who do not require escalation to biologics.
  The higher the percentage of severe asthmatic patients who are escalated to biologics, the worse. The lower the percentage of severe asthmatic patients who are escalated to biologics, the better.
  Change in biologic escalation percentage between baseline, 6-months, and prior published evidence that indicates biologic escalation percentage for those with severe asthma.
  Change in biologic escalation cost will be determined by multiplying the biologic percentage escalation between baseline, 6-months, and prior published evidence by the cost per biologic treatment.
  Cost values will derived either from NHS costing database or published evidence.
Asthma related oral corticosteroids utilization and associated cost | 6 months
  Some patients with asthma who have an exacerbation may require oral corticosteroids. If adherence and technique to a patient's controller inhaled corticosteroid can be improved, there could be less exacerbations and thus, less utilization of oral corticosteroids.
  The higher the percentage of asthmatic patients who are prescribed oral corticosteroids, the worse. The lower the percentage of asthmatic patients who are prescribed oral corticosteroids, the better.
  Change in oral corticosteroid usage for those with asthma will be noted in the 1-year prior to baseline and then from study start to the end of the study.
  Change in oral corticosteroid cost will be determined by multiplying the number of oral corticosteroid doses between 1-year prior to baseline and then from study start to 6-months, by the cost of an oral corticosteroid dose.
  Cost values will derived either from the NHS costing database or published evidence.
Asthma related accident and emergency department visits and associated cost | 6 months
  Some asthma severe exacerbations may require an accident and emergency department visit. If adherence and technique to a patient's controller inhaled corticosteroid can be improved, there could be less exacerbations and thus, less accident and emergency department visits.
  The higher the number of accident and emergency department visits, the worse. The lower the number of accident and emergency department visits, the better.
  Change in accident and emergency department visits will be noted in the 1-year prior to baseline and then from study start to 6-months, the end of the study.
  Change in accident and emergency cost will be determined by multiplying the number of accident and emergency department visits between 1-year prior to baseline and then from study start to 6-months by the cost of an accident and emergency department visit.
  Cost values will derived either from the NHS costing database or published evidence.
Asthma related unscheduled outpatient clinic visits and associated cost | 6 months
  Some patients may have unscheduled outpatient clinic visits due to worsening asthma symptoms or exacerbations. If adherence and technique to controller inhaled corticosteroid is improved, there could be less worsening of symptoms and exacerbations and a decrease in unscheduled outpatient clinic visits.
  The higher the number of unscheduled outpatient clinic visits, the worse. The lower the number of unscheduled outpatient clinic visits, the better.
  Change in unscheduled outpatient clinic visits will be noted in the 1-year prior to baseline and then from study start to 6-months, the end of the study.
  Change in unscheduled outpatient clinic visit cost will be determined by multiplying the number of unscheduled outpatient clinics visits between 1-year prior to baseline and then from study start to 6-months by the cost of an unscheduled outpatient clinic visit.
  Cost values will derived either from the NHS costing database or published evidence.
Asthma related inpatient hospitalization, associated length of stay, and associated cost | 6 months
  Some patients may have asthma related inpatient hospitalizations due to worsening asthma symptoms or exacerbations. If adherence and technique to controller inhaled corticosteroid is improved, there could be less worsening of symptoms and exacerbations and a decrease in inpatient hospitalizations.
  The higher the number of inpatient hospitalizations, the worse. The lower the number of inpatient hospitalizations, the better.
  Change in inpatient hospitalizations will be noted in the 1-year prior to baseline and then from study start to 6-months, the end of the study.
  Change in inpatient hospitalization cost will be determined by multiplying the number of asthma related inpatient hospitalizations between 1-year prior to baseline and then from study start to 6-months by the cost of an inpatient hospitalization.
  Cost values will derived either from the NHS costing database or published evidence.
Computer System Usability Questionnaire | 6 months
  The Computer System Usability Questionnaire is a validated questionnaire that is used in digital health to obtain feedback on the usefulness, ease of use, and satisfaction of digital platform.
  There are 19 questions in the Computer System Usability Questionnaire. Each question has a range between 1 and 7 with 1 = strongly disagree and 7 = strongly agree. For each question, there is an option for not applicable (NA).
  The higher the mean score, the better. The lower the mean score, the worse.
  The Computer System Usability Questionnaire will be administered to all patients at the end of the study.
Semi-structured interviews using the 2019 Rudin et al study | 6 months
  The study by Rudin, R.S., Fanta, C.H., Qureshi, N., Duffy, E., Edelen, M.O., Dalal, A.K., Bates, D.W. (2019). A clinically integrated mHealth app and practice model for collecting patient-reported outcomes between visits for asthma patients: implementation and feasibility. App Clin Inform, 10, 783-793 - contains a validated semi-structured interview used to obtain for feedback on the feasibility, acceptability, and use of digital health technologies. Interviews can be administered to patients and health care providers. There are 7 questions for patients. There are 5 questions for health care providers. There is no score as this is a qualitative survey.
  Interviews will be conducted either in-person or virtually by the clinical research organization, Lindus Health. At the conclusion of the interviews, Lindus Health will then use thematic analysis will be used to determine the main themes.

CONTACTS AND LOCATIONS:
Overall Officials: David J Jackson, MRCP MSc PhD, Principal Investigator — Consultant in Asthma & Eosinophilic Lung Diseases
Locations (1):
- Guy's and St. Thomas' NHS Foundation Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, SAP, ICF, CSR, and all data analyses will be shared by Aptar Digital Health and Lindus Health (our CRO) with the Guy's and St. Thomas' Hospital Severe Asthma Clinical team. This trial has already been approved by the local Research & Ethics Committee.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Barry LE, O'Neill C, Butler C, Chaudhuri R, Heaney LG. Cost-Effectiveness of Fractional Exhaled Nitric Oxide Suppression Testing as an Adherence Screening Tool Among Patients With Difficult-to-Control Asthma. J Allergy Clin Immunol Pract. 2023 Jun;11(6):1796-1804.e3. doi: 10.1016/j.jaip.2023.03.008. Epub 2023 Mar 20. PMID 36940864
- [Result] Boinet T, Leroy-David C. [Asthma in adults]. Actual Pharm. 2021 Feb;60(603):13-17. doi: 10.1016/j.actpha.2020.12.008. Epub 2021 Feb 22. French. PMID 33642669
- [Result] Nordon C, Grimaldi-Bensouda L, Pribil C, Nachbaur G, Amzal B, Thabut G, Marthan R, Aubier M; COBRA Study Group. Clinical and economic burden of severe asthma: A French cohort study. Respir Med. 2018 Nov;144:42-49. doi: 10.1016/j.rmed.2018.10.002. Epub 2018 Oct 2. PMID 30366583
- [Result] Budhathoki P, Shrestha DB, Rawal E, Khadka S. Corticosteroids in COVID-19: Is it Rational? A Systematic Review and Meta-Analysis. SN Compr Clin Med. 2020;2(12):2600-2620. doi: 10.1007/s42399-020-00515-6. Epub 2020 Oct 19. PMID 33103063
- [Result] George M, Bender B. New insights to improve treatment adherence in asthma and COPD. Patient Prefer Adherence. 2019 Jul 31;13:1325-1334. doi: 10.2147/PPA.S209532. eCollection 2019. PMID 31534319
- [Result] Busse WW, Kraft M. Current unmet needs and potential solutions to uncontrolled asthma. Eur Respir Rev. 2022 Jan 25;31(163):210176. doi: 10.1183/16000617.0176-2021. Print 2022 Mar 31. PMID 35082128
- [Result] McDonald VM, Yorke J. Adherence in severe asthma: time to get it right. Eur Respir J. 2017 Dec 21;50(6):1702191. doi: 10.1183/13993003.02191-2017. Print 2017 Dec. No abstract available. PMID 29269587
- [Result] Barnes CB, Ulrik CS. Asthma and adherence to inhaled corticosteroids: current status and future perspectives. Respir Care. 2015 Mar;60(3):455-68. doi: 10.4187/respcare.03200. Epub 2014 Aug 12. PMID 25118311
- [Result] Jackson DJ, Busby J, Pfeffer PE, Menzies-Gow A, Brown T, Gore R, Doherty M, Mansur AH, Message S, Niven R, Patel M, Heaney LG; UK Severe Asthma Registry. Characterisation of patients with severe asthma in the UK Severe Asthma Registry in the biologic era. Thorax. 2021 Mar;76(3):220-227. doi: 10.1136/thoraxjnl-2020-215168. Epub 2020 Dec 9. PMID 33298582
- [Result] Blakey JD, Bender BG, Dima AL, Weinman J, Safioti G, Costello RW. Digital technologies and adherence in respiratory diseases: the road ahead. Eur Respir J. 2018 Nov 22;52(5):1801147. doi: 10.1183/13993003.01147-2018. Print 2018 Nov. PMID 30409819
- [Result] Merchant R, Szefler SJ, Bender BG, Tuffli M, Barrett MA, Gondalia R, Kaye L, Van Sickle D, Stempel DA. Impact of a digital health intervention on asthma resource utilization. World Allergy Organ J. 2018 Dec 3;11(1):28. doi: 10.1186/s40413-018-0209-0. eCollection 2018. PMID 30524644
- [Result] Chan A, De Simoni A, Wileman V, Holliday L, Newby CJ, Chisari C, Ali S, Zhu N, Padakanti P, Pinprachanan V, Ting V, Griffiths CJ. Digital interventions to improve adherence to maintenance medication in asthma. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD013030. doi: 10.1002/14651858.CD013030.pub2. PMID 35691614
- [Result] Lara M, Edelen MO, Eberhart NK, Stucky BD, Sherbourne CD. Development and validation of the RAND Asthma Control Measure. Eur Respir J. 2014 Nov;44(5):1243-52. doi: 10.1183/09031936.00051614. Epub 2014 Jul 17. PMID 25034567
- [Result] Sherbourne CD, Stucky BD, Edelen MO, Eberhart NK, Kleerup E, Lara M. Assessing the validity of the RAND negative impact of asthma on quality of life short forms. J Allergy Clin Immunol. 2014 Oct;134(4):900-7. doi: 10.1016/j.jaci.2014.03.002. Epub 2014 Apr 18. PMID 24746752
- [Result] Rudin RS, Fanta CH, Qureshi N, Duffy E, Edelen MO, Dalal AK, Bates DW. A Clinically Integrated mHealth App and Practice Model for Collecting Patient-Reported Outcomes between Visits for Asthma Patients: Implementation and Feasibility. Appl Clin Inform. 2019 Oct;10(5):783-793. doi: 10.1055/s-0039-1697597. Epub 2019 Oct 16. PMID 31618782
- See also: Global Initiative for Asthma (GINA). Global Strategy for Asthma Management and Prevention, 2022. — https://www.ginasthma.org
- See also: World Health Organization (WHO). Asthma. 12 May 2022. — https://www.who.int/news-room/fact-sheets/detail/asthma
- See also: American Academy of Pediatrics. (2022). Mild, moderate, severe asthma: what do grades mean? — https://www.healthychildren.org/English/health-issues/conditions/allergies-asthma/Pages/Mild-Moderate-Severe-Asthma-What-Do-Grades-Mean.aspx
- See also: NICE. Asthma: diagnosis, monitoring, and chronic asthma management. NICE guideline NG80. March 22, 2021. — http://www.nice.org.uk/guidance/ng80
- See also: NICE. Medicines adherence: involving patients in decisions about prescribed medicines and supporting adherence. NICE guidance CG76. January 28, 2009. — http://www.nice.org.uk/guidance/cg76
- See also: NICE. Measuring fractional exhaled nitric oxide concentration in asthma: NIOX MINO, NIOX VERO, and NObreath. NICE guidance DG12. April 2, 2014. — http://www.nice.org.uk/guidance/dg12
- See also: Oxford Academic Health Science Network. Consensus pathway for management of uncontrolled asthma in adults. June 2022. — https://www.oxfordahsn.org/our-work/asthma-biologics-toolkit/aac-consensus-pathway-for-management-of-uncontrolled-asthma-in-adults/